CLINICAL TRIAL: NCT02945436
Title: Optimizing HIV Counseling and Testing and Referral Through an Adaptive Drug Use
Brief Title: Optimizing HIV Counseling and Testing and Referral Through an Adaptive Drug Use Intervention
Acronym: Swerve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Robert Stephenson, Professor, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: HUM00105125; R01DA041032-02 (NIH)
Record Dates: First submitted 2016-10-17; First posted 2016-10-26 (Estimated); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: HIV; Substance Use
MeSH Terms: conditions — Substance-Related Disorders | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SOC + SOC (Active Comparator): Participants will receive current standard of care (SOC) for HIV counseling, testing, and referral at both visit 1 and visit 2.
  Interventions: Behavioral: Standard of Care (SOC)
- SOC + SUBI (Experimental): Participants will receive SOC at visit 1 and the experimental substance use brief intervention (SUBI) at visit 2.
  Interventions: Behavioral: Substance Use Brief Intervention; Behavioral: Standard of Care (SOC)
- SUBI + SUBI (Experimental): Participants will receive the SUBI at both visit 1 and visit 2.
  Interventions: Behavioral: Substance Use Brief Intervention
- SUBI + SOC (Experimental): Participants will receive the SUBI at visit 1 and SOC at visit 2.
  Interventions: Behavioral: Substance Use Brief Intervention; Behavioral: Standard of Care (SOC)

INTERVENTIONS:
Behavioral: Substance Use Brief Intervention — SUBI is a counseling intervention based on Motivational Interviewing techniques that focuses on the substance use and sexual health risks of participants.
  Other Names: SUBI
  Arms: SOC + SUBI; SUBI + SOC; SUBI + SUBI
Behavioral: Standard of Care (SOC) — Standard of care is Counseling Testing and Referral (CTR). CTR is a standardized service in which counselors provide HIV testing, risk-related counseling and appropriate referrals (medical, social, prevention, and partner services) to clients.
  Arms: SOC + SOC; SOC + SUBI; SUBI + SOC

SUMMARY:
A sample of 300 young (15-29) men who have sex with men (MSM) and transgender persons living in South-East Michigan's Detroit Metro Area (DMA) will be recruited through venue-based sampling and online ads to examine the efficacy of adding a substance use brief intervention (SUBI) to standard HIV prevention and care (SOC) for achieving gains in successful engagement in HIV care. The investigators will partner with Detroit-area AIDS Service Organizations (ASOs) to deliver the intervention.

DETAILED DESCRIPTION:
The research activities involve a prospective 4-arm factorial RCT (SOC-only, SOC+SUBI, SUBI+SOC, SUBI+SUBI) of approximately 300 ATOD-using high-risk YMSM aged 15-29 in the DMA. The intervention comprises of two intervention visits, at which time participants may get either standard of care only (SOC-only) or standard of care plus SUBI. All participants will receive standard of care (SOC; i.e., Comprehensive HIV Testing and Counseling) at each visit. The substance use brief intervention (SUBI) will be added to SOC within the experimental arms. At intervention visit one, standard of care is the same for all participants: standard of care is Counseling Testing and Referral (CTR).CTR is a standardized service in which counselors provide HIV testing, risk-related counseling and appropriate referrals (medical, social, prevention, and partner services) to clients. Hence at visit one, 150 YMSM will receive CTR and 150 YMSM will receive CTR+SUBI. The investigators expect approximately 10-15% of participants to test HIV positive at intervention visit one. For intervention visit two, standard of care is sero-status specific. For HIV-negatives standard of care remains CTR. For HIV-positives standard of care is case management, as offered routinely by each ASO, which involves counseling on linkage to care and the importance of care retention. To examine how the sequencing and dosing of interventions impacts efficacy, the investigators propose to randomize at baseline into a factorial randomized controlled trial. The control arm will receive SOC-only at both intervention visit one and two (SOC-only). Experimental arm one (SOC+SUBI) will receive SOC at visit one and SUBI at visit two. Experimental arm two (SUBI+SOC) will receive SUBI at visit one and SOC at visit two. Experimental arm three (SUBI+SUBI) will receive the intervention condition at visits one and two.

The RCT thus answers two important questions: 1) What is the impact of the addition of SUBI to SOC on HIV engagement in care and sexual and substance-related risk-taking behaviors among high-risk YMSM? and 2) What combination of services (SOC-only, SOC+SUBI, SUBI+SOC, SUBI+SUBI) has the greatest impact on engagement in HIV prevention? (where engagement in care is defined as routine HIV testing for sero-negative YMSM and linkage/retention in care for sero-positive MSM).

ELIGIBILITY:
Inclusion Criteria:

* All participants must be ages 15-29
* All participants must currently reside in the DMA (verified by zip code)
* All participants must self-report as HIV sero-negative
* All participants must report at least one sexual experience with a man in the previous 6 months
* All participants must report either at least one binge-drinking episode and/or use of illicit substances in the previous 3 months
* All participants must identify as either a man who has sex with men (MSM) or as transgender
* All participants must speak English

Exclusion Criteria:

°Anyone not meeting all 6 inclusion criteria will be excluded from the study

Ages: 15 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 258 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Increases in repeat HIV testing | 18 months
  Increases in repeat HIV testing as measured by the "HIV Testing Questions" section of the questionnaires

OTHER OUTCOMES:
Decreases in sexual risk behavior | 18 months
  Decreases in sexual risk behavior as measured by the "Sexual History" section of the questionnaires
Reduction in substance use and abuse as measured by the "Assist", "Audit", "Medical Marijuana", Synthetic Cannabis", "Energy Drinks", and "Substance Use (past 30 days)" sections of the questionnaires | 18 months
  Investigators will verify self-reported substance use by collecting and testing biological samples. Investigators will measure alcohol use with an Ethyl Glucuronide (ETG) urine test. Investigators will measure the use of other substances with an EZ Split Key Cup urine test.
Reduction in consequences of substance use as measured by the "Assist", "Audit" and "Overdose" sections of the questionnaires | 18 months
  Reduction in the number of participants who experience negative consequences of substance use as measured by the "Assist", "Audit" and "Overdose" sections of the questionnaires
Decreased STI incidence | 18 months
  Decreases in STI incidence as measured by the "STI History" section of the questionnaires
Increase in the number of participants who have been successfully engaged in care | 18 months
  The investigators define engagement in HIV care as linkage and retention in HIV care (per the Institute of Medicine guidelines of linkage, or first HIV-care related visit, within 90 days of diagnosis and at least two physician visits with a CD4 and viral load test in 12 months) and achievement of viral suppression.

CONTACTS AND LOCATIONS:
Overall Officials: Rob Stephenson, PhD, Principal Investigator — Director, Professor
Locations (1):
- Center for Sexuality and Health Disparities, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parker JN, Choi SK, Bauermeister JA, Bonar EE, Carrico AW, Stephenson R. HIV and Sexually Transmitted Infection Testing Among Substance-Using Sexual and Gender Minority Adolescents and Young Adults: Baseline Survey of a Randomized Controlled Trial. JMIR Public Health Surveill. 2022 Jul 1;8(7):e30944. doi: 10.2196/30944. PMID 35776441
- [Derived] Parker JN, Hunter AS, Bauermeister JA, Bonar EE, Carrico A, Stephenson R. Comparing Social Media and In-Person Recruitment: Lessons Learned From Recruiting Substance-Using, Sexual and Gender Minority Adolescents and Young Adults for a Randomized Control Trial. JMIR Public Health Surveill. 2021 Dec 1;7(12):e31657. doi: 10.2196/31657. PMID 34855613
- [Derived] Stephenson R, Bonar EE, Carrico A, Hunter A, Connochie D, Himmelstein R, Bauermeister J. Intervention to Increase HIV Testing Among Substance-Using Young Men Who Have Sex With Men: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2018 Apr 30;7(4):e114. doi: 10.2196/resprot.9414. PMID 29712625